CLINICAL TRIAL: NCT04265378
Title: Effects of Cognitive Training and Brain Stimulation in Prodromal Alzheimer's Disease - Randomised, Sham Controlled, Interventional Study
Brief Title: Cognitive Training and Brain Stimulation in Prodromal Alzheimer's Disease
Acronym: AD-Stim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-Stim
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Subjective Cognitive Decline; Mild Cognitive Impairment
Keywords: memory; brain stimulation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimulation group (Experimental): Anodal tDCS + intensive cognitive training
  Interventions: Device: anodal tDCS; Behavioral: Intensive cognitive training
- Sham group (Sham Comparator): Sham tDCS + intensive cognitive training
  Interventions: Behavioral: Intensive cognitive training

INTERVENTIONS:
Device: anodal tDCS — Anodal transcranial direct current stimulation (tDCS), 9 sessions with 20 minutes stimulation each (current intensity of 1mA)
  Arms: Stimulation group
Behavioral: Intensive cognitive training — Intensive cognitive training of a letter memory updating task and a 3-stage Markov decision making task, 9 sessions

SUMMARY:
The aim of this study is to investigate whether a tDCS-accompanied intensive cognitive training of working memory leads to performance improvement in individuals with prodromal Alzheimer's disease.

DETAILED DESCRIPTION:
The goal of the present study is to assess behavioral (primary) effects of a multi-session cognitive training combined with transcranial direct current stimulation (tDCS). Many studies to date have found tDCS to be an efficient method to enhance various cognitive functions by modulating cortical excitability in young adults, but its behavioral impact and underlying mechanisms in pathological aging still need to be elucidated. Individuals with prodromal Alzheimer's disease, will participate in a three-week cognitive training with concurrent online tDCS application. Cognitive performance (primary) will be examined before, during and after the intervention, in order to draw conclusions about the effect of tDCS. In addition to cognitive training, a control group, receiving sham stimulation during training, will be assessed. Follow-up sessions to assess long-term effects are planned four weeks and seven months after the post assessment. Furthermore, to assess potential predictors of tDCS effects, functional and structural parameters will be measured with MRI. The results of the study will offer valuable insights into efficacy of combined tDCS and cognitive training, as compared to training alone, in individuals with prodromal stages of Alzheimer's disease. Moreover, improved understanding of tDCS effects on cognitive training performance and underlying neural correlates may help to develop novel approaches for modulating cognitive decline in healthy and pathological aging.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (60 - 80 years);
* Right handedness;
* subjective cognitive decline (SCD) or mild cognitive impairment (MCI)

Exclusion Criteria:

* Dementia or other neurodegenerative neurological disorders; epilepsy or history of seizures; close relatives with epilepsy or history of seizures; previous stroke;
* Severe and untreated medical conditions that precludes participation in the training, as determined by responsible physician;
* History of severe alcoholism or use of drugs;
* Severe psychiatric disorders such as depression (if not in remission) or psychosis

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Working memory training performance (Letter Updating task) | 3 weeks
  Performance in a memory training task (Letter updating) under anodal tDCS compared to sham condition; operationalized by working Memory Updating performance assessed with number of correctly recalled letter lists in the letter updating task, analyzed immediately after training period (anodal condition versus sham)

SECONDARY OUTCOMES:
Working memory training performance (Markov task) | 3 weeks
  Performance in second memory training task (Markov decision making) under anodal tDCS compared to sham condition, analyzed immediately after training period (anodal condition versus sham)
Transfer outcomes: numerical n-back task (% correct) | 3 weeks
  Comparing performance immediately before and after training period (anodal condition versus sham)
Transfer outcomes: AVLT (auditory verbal learning test) (sum of correctly recalled items trials 1-5) | 3 weeks
  Comparing performance immediately before and after training period (anodal condition versus sham)
Transfer outcomes: Wiener Matrices Test (no. correct) | 3 weeks
  Comparing performance immediately before and after training period (anodal condition versus sham)
Long-term outcomes: Letter Updating task (no. of correctly recalled lists) | 4 weeks and 7 months after training
  Comparing performance immediately before and after training period with performance at 4 weeks and 7-months after training period (anodal condition versus sham)
Long-term outcomes: Markov decision making task (% optimal actions) | 4 weeks and 7 months after training
  Comparing performance immediately before and after training period with performance at 4 weeks and 7-months after training period (anodal condition versus sham)
Long-term outcomes: numerical n-back task (% correct) | 4 weeks and 7 months after training
  Comparing performance immediately before and after training period with performance at 4 weeks and 7-months after training period (anodal condition versus sham)
Long-term outcomes: AVLT (auditory verbal learning test) (sum of correctly recalled items trials 1-5) | 4 weeks and 7 months after training
  Comparing performance immediately before and after training period with performance at 4 weeks and 7-months after training period (anodal condition versus sham)
Long-term outcomes: Wiener Matrices Test (no. correct) | 4 weeks and 7 months after training
  Comparing performance immediately before and after training period with performance at 4 weeks and 7-months after training period (anodal condition versus sham)
Neural correlates: Structural neural correlates of tDCS effect | before training; 7 months after training
  - structural neural correlates; assessed by grey matter volumes, cortical thickness, white matter microstructure (diffusion tensor imaging (DTI) measures: fractional anisotropy, mean diffusivity)
  before the intervention and at 7-months after training period (correlations in anodal group)
Neural correlates: Functional neural correlates of tDCS effect | before training; 7 months after training
  - functional neural correlates; assessed by resting-state fMRI analyses to obtain functional connectivities (seed-based connectivity: correlation of BOLD-timeseries between a seed/ROI and every voxel/location in the brain)
  before the intervention and at 7-months after training period (correlations in anodal group)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antonenko D, Fromm AE, Thams F, Kuzmina A, Backhaus M, Knochenhauer E, Li SC, Grittner U, Floel A. Cognitive training and brain stimulation in patients with cognitive impairment: a randomized controlled trial. Alzheimers Res Ther. 2024 Jan 11;16(1):6. doi: 10.1186/s13195-024-01381-3. PMID 38212815
- [Derived] Thams F, Kuzmina A, Backhaus M, Li SC, Grittner U, Antonenko D, Floel A. Cognitive training and brain stimulation in prodromal Alzheimer's disease (AD-Stim)-study protocol for a double-blind randomized controlled phase IIb (monocenter) trial. Alzheimers Res Ther. 2020 Nov 7;12(1):142. doi: 10.1186/s13195-020-00692-5. PMID 33160420

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT04265378/SAP_001.pdf